CLINICAL TRIAL: NCT06818422
Title: Comparison of Telemedicine and Conventional Monitoring Methods in Nonspecific Neck Pain
Brief Title: Telemedicine for Nonspecific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Antalya EAH, Antalya ŞH
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain; Exercise; Telemedicine
Keywords: neck pain; home exercise; telemedicine; teleexercise
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of the procedures used in the other group. Additionally, the outcome assessor will be blinded to group assignments during the statistical analysis to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine Group (Experimental): Patients will receive pre-recorded neck exercise and educational videos sent to their phones by the physician. They will follow the exercise routine at home three times a day for 2 weeks, based on the provided videos. They will mark the exercise diary given to them when they do their exercises. They will be advised to continue exercise program for 3 months. Additionally, the physician will conduct video calls to monitor their pain levels and offer support at the 15th day, 30th day and the 3rd month of the study.
  Interventions: Other: Home exercise and recommendations for nonspecific neck pain
- Conventional Follow-up Group (Active Comparator): Patients will receive an exercise brochure and a brochure with educational recommendations given by a physician face-to-face in the clinic. These patients will follow the exercise routine at home three times a day for 2 weeks, based on the provided brochures. They will mark the exercise diary given to them when they do their exercises. They will also be advised to continue exercises for 3 months. They will be come to clinic check-ups to monitor pain intensity and provide support at the 15th day, 30th day and the 3rd month of the study.
  Interventions: Other: Home exercise and recommendations for nonspecific neck pain

INTERVENTIONS:
Other: Home exercise and recommendations for nonspecific neck pain — The intervention involves neck exercises and recommendations for nonspecific neck pain. Patients will perform the exercises at home three times a day for 2 weeks and record their progress in an exercise diary. They will be monitored by a physician for pain levels and receive additional support at the 15th day, 30th day and 3rd months.

SUMMARY:
Brief Summary

Neck pain is a common global health issue, often classified as nonspecific neck pain when no specific cause is identified. This study aims to compare the effectiveness of telemedicine (which involves providing home exercises and recommendations through pre-recorded exercise videos and remote follow-up) versus conventional care (which involves providing home exercises and recommendations through informational brochures and in-person follow-ups) for patients with nonspecific neck pain. Participants will be randomly assigned to either group. The primary outcomes are pain intensity (VAS) and neck function (NDI), with secondary outcomes including exercise adherence, patient satisfaction, and time and distance spent for in-patient follow-ups.

The study hypothesizes that telemedicine will result in greater pain reduction, improved neck function, and higher patient satisfaction due to the convenience and accessibility of video-based exercises. If proven effective, telemedicine could reduce hospital crowding, minimize infection risks, save time and money, and reduce environmental impacts, making it a valuable tool in non-serious pathologies and during events like pandemics.

DETAILED DESCRIPTION:
Neck pain is a very common public health problem worldwide. It is defined as pain perceived between the upper nuchal line and the spinous process of the first thoracic vertebra. This pain can sometimes be reflected to the head, trunk and upper extremities. Nonspecific neck pain refers to neck pain for which no specific cause or underlying disease can be identified. It is generally used to refer to neck pain that cannot be attributed to conditions such as infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder or radicular symptoms. Although many interventions have been recommended for neck pain in the American Physical Therapy Association (APTA) clinical practice guideline, the only interventions recommended based on strong evidence are coordination, strengthening, endurance exercises, cervical mobilization/manipulation and patient education. Other interventions are based on weak or moderate evidence. In neck pain syndromes, exercise therapy is primarily recommended for neck pain without signs of major structural pathology. In fact, exercise therapy has surpassed physical therapy modalities compared to the past. While exercise, mobilization, and manipulation treatments for non-specific neck pain have the greatest support in the literature, there is little evidence for the effectiveness of thermal treatments and electrical therapies, with no evidence of more than a temporary benefit.

This study aims to compare the telemedicine method, in which asynchronous exercise videos (tele-exercise) and educational videos containing recommendations (tele-education) are sent to patients' phones, and patients are followed up by physicians via remote video calls (tele-consultation), with the conventional follow-up method, in which patients are given a brochure containing the same exercises and recommendations, and patients are followed up by physicians via face-to-face meetings in the hospital.

Participants will consist of patients diagnosed with non-specific neck pain for at least 3 months. Patients will be randomly assigned to one of two groups: Group A (Telemedicine Group) and Group B (Conventional Follow-up Group). The study content will be explained to the patients on the first day at the hospital and they will be asked to sign a voluntary consent form. Patients in Group A will receive a pre-recorded neck exercise video and an educational video sent to their phones by the physician. These patients will exercise at home three times a day for 3 months. They were told to mark the exercise diary provided to them when they do their exercises for 2 weeks. They will have remote check-ups via video call on the 15th day, 30th day and 3rd month to monitor pain intensity and provide support. Patients in Group B will receive an exercise brochure and an educational brochure provided by the physician in person at the clinic. These patients will also be advised to exercise at home three times a day for 3 months. For 2 weeks period they were told to mark the exercise diary provided to them when they do their exercises. They will have clinical check-ups on the 15th day, 30th day and 3rd month to monitor pain intensity and provide support. The primary outcome measures are pain intensity measured using the Visual Analog Scale (VAS) and neck function assessed using the Neck Disability Index (NDI). Secondary outcome measures are adherence to the exercise program monitored through an exercise diary, patient satisfaction assessed on a Likert scale from 0 to 5, and distance in kilometers and time in hours or minutes (spent on the road to hospital) for Group B.

VAS and NDI will be measured initially for both groups through face-to-face assessments, and total distance and time spent on transportation will be calculated for Group B. In 15th day, VAS will be administered through video interviews (Group A) and face-to-face assessments (Group B). In addition, completed exercise diaries will be collected via WhatsApp (Group A) or clinic visits (Group B). In 30th day, VAS and in 3rd month VAS, NDI and patient satisfaction will be assessed through video interviews (Group A) and face-to-face assessments (Group B).

Participants will be unaware of the procedures used in the other group and the outcome assessor will be blinded to group assignments during the statistical analysis to prevent bias. Adherence will be monitored through exercise diaries and qualitative feedback will be collected through surveys or interviews to understand patient experiences and compliance difficulties. Sample size will be determined based on power analysis.

The primary hypothesis (H1) is that Group A will show greater improvement in pain reduction and neck function than Group B due to the more accurate implementation of video exercises and advice than visual exercises and advice. The secondary hypothesis (H2) is that Group A will show higher adherence and satisfaction due to the ease of video-based exercises and the lack of a hospital visit.

This study will be the first scientific study to compare the telemedicine method with the conventional method. If the telemedicine method shows an effectiveness this method can be widely used in the future, this will provide great convenience for both clinicians and patients, reduce the density in hospital polyclinics and reduce the risk of contamination in healthcare areas. Telemedicine applications that can be performed remotely in diseases that do not involve serious pathology provide significant advantages to both individuals and health insurance systems in terms of time (time spent on the road, waiting time in the hospital, etc.) and financial expenses (transportation and healthcare expenses, etc.). In addition, these methods reduce air pollution by reducing traffic density and gasoline consumption, thus minimizing environmental impacts. The spread of telemedicine applications also stands out as an effective medical option in unexpected quarantine conditions such as pandemics.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain for at least 3 months (neck pain without a specific underlying cause such as infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder or radicular symptoms)
* Clinical and/or radiological presence of one of the following diagnoses: cervicalgia, cervical flattening, cervical arthrosis, cervical discopathy
* Able to understand and apply the given exercises; literate and therefore able to read and interpret the given brochure; familiar with smartphones, tablets and computers, able to use them easily, able to open and watch sent videos, have internet access

Exclusion Criteria:

* Having a cognitive disorder
* Red flag findings indicating serious pathology, recent trauma to the neck region, fracture, lysis, listhesis, spinal mass and malignancy, syringomyelia, presence of canal stenosis
* Having undergone surgery in the cervical region
* Having received injections to the neck and back region in the last 3 months
* Having received physical therapy or home exercise recommendations in the same hospital or in another center in the last 3 months
* Not having their own smartphone or smart tablet and/or uninterrupted internet access
* Having a visual impairment
* Having an upper extremity amputation
* Having advanced cancer, receiving cancer treatment
* Having complicated diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline, 15th day, 30th day and 3rd month
  Pain intensity will be measured using the Visual Analog Scale (VAS). Minimum value is 0 (no pain), maximum value is 10 (most imaginable pain).
Neck function | Baseline and 3rd month
  Neck function will be assessed using the Neck Disability Index (NDI). Minimum value is 0 (no disability), maximum value is 50 (maximum disability).

SECONDARY OUTCOMES:
Adherence to the exercise program | 15th day
  Adherence to the exercise program will be evaluated by reviewing the exercise diaries completed by the patients. This assessment will allow us to gauge their compliance and overall performance in the program. the patients. We will review these diaries to evaluate their compliance.
Patient satisfaction | 3rd month
  Patient satisfaction will be assessed using a Likert scale from 0 to 5.
Transportation distance | Baseline
  Total distance (km) necessary to go to follow-up visits will be asked and noted for group B.
The time spent | Baseline
  Total time (hours/minutes) spent for follow-up visits will be recorded for Group B.

CONTACTS AND LOCATIONS:
Overall Officials: Selkin Yılmaz Muluk, MD, Principal Investigator — Antalya Training and Research Hospital, Antalya City Hospital
Locations (3):
- Turkey (Türkiye) (3):
  - Selkin Yılmaz Muluk, Antalya
  - Antalya City Hospital, Antalya
  - Antalya Training and Research Hospital, Antalya

IPD SHARING:
Plan to Share IPD: Yes
I am planning to share a portion of the study plan, specifically the plan description section, with the public. This will provide transparency and allow for greater engagement with the community regarding our research objectives and methodology.
Supporting Information: Study Protocol
Time Frame: I plan to share the study protocol with the public once it has received the necessary approvals from the relevant authorities.
Access Criteria: Access to the study protocol will be granted to individuals and organizations interested in our research, subject to the approval of the relevant ethical and regulatory bodies. This includes researchers, healthcare professionals, and members of the public who seek to understand the study's objectives and methodology

REFERENCES:
- [Background] Fandim JV, Nitzsche R, Michaleff ZA, Pena Costa LO, Saragiotto B. The contemporary management of neck pain in adults. Pain Manag. 2021 Jan;11(1):75-87. doi: 10.2217/pmt-2020-0046. Epub 2020 Nov 25. PMID 33234017
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Guzman J, Hurwitz EL, Carroll LJ, Haldeman S, Cote P, Carragee EJ, Peloso PM, van der Velde G, Holm LW, Hogg-Johnson S, Nordin M, Cassidy JD. A new conceptual model of neck pain: linking onset, course, and care: the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S17-28. doi: 10.1016/j.jmpt.2008.11.007. PMID 19251062
- [Background] Bier JD, Scholten-Peeters WGM, Staal JB, Pool J, van Tulder MW, Beekman E, Knoop J, Meerhoff G, Verhagen AP. Clinical Practice Guideline for Physical Therapy Assessment and Treatment in Patients With Nonspecific Neck Pain. Phys Ther. 2018 Mar 1;98(3):162-171. doi: 10.1093/ptj/pzx118. PMID 29228289
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Swenson RS. Therapeutic modalities in the management of nonspecific neck pain. Phys Med Rehabil Clin N Am. 2003 Aug;14(3):605-27. doi: 10.1016/s1047-9651(03)00038-x. PMID 12948344
- See also: Neck exercises — http://www.oxfordhealth.nhs.uk
- See also: Neck exercises — http://www.csp.org.uk
- See also: Neck exercises — http://www.nhs.uk